CLINICAL TRIAL: NCT04132843
Title: Novel Multi-Parameter Mapping and Analysis Techniques for Characterization and Treatment Assessment of High Grade Brain Lesions
Brief Title: Novel MRI Techniques for the Characterization and Treatment Assessment of High Grade Brain Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0324; NCI-2019-05781 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0324 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-09-05; First posted 2019-10-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Brain Neoplasm; Lymphoma; Metastatic Malignant Neoplasm in the Brain; Recurrent Malignant Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Lymphoma | interventions — gadobenic acid; gadobutrol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (MRI, gadobutrol, gadobenate dimeglumine) (Experimental): Within 21 days before standard of care chemotherapy and/or radiation therapy, patients undergo an MRI scan for the first set of images. Patients then receive either gadobutrol or gadobenate dimeglumine IV and undergo an MRI for the second set of images. All MRI scans take a total of 60 minutes to complete. Patients then repeat the MRI scans 120 days after standard of care chemotherapy and/or radiation therapy.
  Interventions: Drug: Gadobenate Dimeglumine; Drug: Gadobutrol; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Gadobenate Dimeglumine — Given IV
  Other Names: Gd-BOPTA; MultiHance
Drug: Gadobutrol — Given IV
  Other Names: BAY86-4875; Gadavist; Gadograf; Gadovist; Protovis; ZK 135079
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This trial studies different magnetic resonance imaging (MRI) techniques and their ability to provide clearer pictures of lesions in patients with high grade brain lesions. An MRI is a type of imaging scan. Using different MRI techniques to produce clearer images of the brain may help researchers learn about the features of brain lesions and the effects of chemotherapy and/or radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To use 3-dimensional (3D) quantitative mapping to determine whether differences in T2 spin parameters exist between the peritumoral area and normal brain in the contralateral hemisphere at baseline.

II. To use 3D quantitative mapping to examine how differences between peritumoral and normal brain in the contralateral hemisphere change before and after treatment.

SECONDARY OBJECTIVES:

I. Determine whether T2 values might be useful in distinguishing non-enhancing components of the tumor as well as predicting response to treatment.

II. Quantify T1 and proton density (PD) spin parameters of the peritumoral area and their differences before and after treatment.

III. Examine post-contrast T1 spin parameters with perfusion characteristics as measured by an established dynamic susceptibility contrast (DSC) technique.

IV. Examine differences in measured perfusion parameters (blood volume and mean transit time of each tumor) before and after treatment.

OUTLINE:

Within 21 days before standard of care chemotherapy and/or radiation therapy, patients undergo an MRI scan for the first set of images. Patients then receive either gadobutrol or gadobenate dimeglumine intravenously (IV) and undergo an MRI for the second set of images. All MRI scans take a total of 60 minutes to complete. Patients then repeat the MRI scans 120 days after standard of care chemotherapy and/or radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least one enhancing lesion, aggregate of enhancing foci, and nonenhancing lesion measuring at least 1 cm in size and is suspected to be a high grade brain neoplasm
* Patient is dispositioned to surgery, chemotherapy and/or radiation therapy
* Patient is able to understand and give own consent to participate in the study

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI) as assessed by our standard of care magnetic resonance (MR) screening procedure, which includes implants or devices that are unsafe in the magnetic environment
* Contraindication or history of allergy to Gadolinium-based (gadobutrol [Gadovist], gadobenate dimeglumine (Multihance]) intravenous contrast
* Verbal confirmation of pregnancy or a positive pregnancy test result in patient record
* Prior partial (greater than 50%) or gross total resection of primary tumor
* Prior chemotherapy or radiation treatment to brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Differences in T2 spin parameters | Baseline
  Will use 3-dimensional (3D) quantitative mapping to determine whether different in T2 spin parameters exist between the peritumoral area and normal brain in the contralateral hemisphere. If the data are normal, will calculate 95% confidence intervals around the mean paired difference in baseline T2 between the peritumoral and normal regions. If the data are not normally distributed, ordered statistics will be calculated, and bootstrapping will be used to estimate the 2.5th and 97.5th percentiles for the median.
Differences between peritumoral and normal brain | Baseline up to 120 days
  Will use 3D quantitative mapping to examine how differences between peritumoral and normal brain in the contralateral hemisphere change before and after treatment. The regions of interest drawn on measured magnetic resonance (MR) spin parameter and MR perfusion parameter values will be grouped according to time point (pre- or post-treatment) and area (peritumoral, tumoral, and normal brain in the contralateral hemisphere). Descriptive statistics and boxplots of these measurements, paired differences between areas and paired differences between time points will be calculated. Will calculate 95% confidence intervals around the mean paired change between area differences at baseline and post-treatment.

SECONDARY OUTCOMES:
Usefulness of T2 values in distinguishing non-enhancing components of the tumor | Up to 120 days
  Will use area under an receive operating curve to determine whether T2 values might be useful in distinguishing non-enhancing components of the tumor as well as predicting response to treatment. Paired data from all patients will be used in this analysis.
Quantification of T1 and proton density (PD) parameters | Baseline up to 120 days
  Will quantify T1 and PD spin parameters of the peritumoral area and their differences before and after treatment.
Post-contrast T1 spin parameters with perfusion characteristics | Up to 120 days
  Will examine post-contrast T1 spin parameters with perfusion characteristics as measured by an established dynamic susceptibility contrast technique.
Differences in measured perfusion parameters before and after treatment. | Baseline up to 120 days
  Will examine differences in measured perfusion parameters before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ken-Pin Hwang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org